CLINICAL TRIAL: NCT06744335
Title: Prospective Observational Multicenter Study of Patients With Arterial Hypertension and Chronic Kidney Disease Markers in Kazakhstan (PROGRESS-CKD)
Brief Title: Prospective Observational Multicenter Study of Patients With AH and CKD Markers in Kazakhstan (PROGRESS-CKD)
Acronym: D1843R00359
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00359
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rate of CKD Diagnosis in Patients With AH and CKD Markers; Demographic and Clinical Characteristics for Those Patients; Routine Therapy Before and After the Diagnosis of CKD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Multicenter, non-interventional PRospective Observational study with retrospective analysis to describe the rate of CKD diaGnosis in patients with aRtErial hypErtenSion and CKD markerS in Kazakhstan

DETAILED DESCRIPTION:
Primary endpoints:

The proportion of patients with markers of chronic kidney disease (CKD) among patients with arterial hypertension such as: albuminuria/proteinuria; GFR <60 ml/min/1.73 m2 (CFR categories C3a-C5).

Secondary endpoints:

The following secondary endpoints will be evaluated in all patients with AH and markers of CKD included in the study (Full Analysis Sampling - FAS) (Secondary Aim 1) and in the subgroup of patients with a diagnosis of CKD confirmed during the study (Modified Full Analysis Sampling - mFAS), i.e., at Visit 1 or

Visit 2 (Secondary Aim 2):

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years at the time of inclusion;

* Patient signed and dated written informed consent form (ICF) in accordance with ICH GCP and local legislation prior to inclusion in the study for the prospective observational cohort;
* Established diagnosis of hypertension, diagnosed in accordance with current clinical guidelines for hypertension, i.e. in adults, i.e. systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg. when measured at two different visits
* Laboratory markers of CKD (eGFR <60 mL/min/1.73 m2 and/or albuminuria/proteinuria*) measured during the period ≤12 months prior to inclusion in the study and persisting ≥3 months between two measurements without a recorded diagnosis of CKD in the primary medical record prior to inclusion;

  * any of the following: urine albumin/creatinine ratio (UACR) ≥30 mg/g (3 mg/mmol), Urine protein-creatinine ratio (uPCR) ≥150 mg/g (15 mg/mmol), albuminuria ≥30 mg/d or Urine protein-creatinine ratio (uPCR) ≥0.15 mg/d.
* Absence of documented diagnosis of CKD in the patient's medical records prior to inclusion in the study

Exclusion Criteria:

* Absence of a signed ICF in patients in the prospective follow-up group

  * Participation in any randomized controlled trial within 3 months prior to inclusion in this study or during participation in this study
  * An established diagnosis of type 1 or type 2 diabetes mellitus.
  * Diagnosis of symptomatic chronic heart failure (CHF), NYHA functional class III-IV, documented in the patient's medical records
  * Diagnosis of AH of secondary genesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned study population for the prospective analysis consists of 1,282 adult outpatients with AH with one or more markers of CKD, without a documented diagnosis of CKD before inclusion in the study and without a documented diagnosis of DM or III-IV stage chronic heart failure (CHF). The planned number of study centers is ~15 outpatient sites in approximately 10 regions of Kazakhstan.
  The retrospective part includes a physician's retrospective review of the ambulatory cards or medical records of outpatients with a reported diagnosis of arterial hypertension for the presence of laboratory markers of CKD assessed ≥3 and ≤12 months prior to inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1282 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with markers of chronic kidney disease (CKD) among patients with arterial hypertension such as: albuminuria/proteinuria; GFR <60 ml/min/1.73 m2 (CFR categories C3a-C5). | 16 months
  The proportion of patients with markers of chronic kidney disease (CKD) among patients with arterial hypertension such as: albuminuria/proteinuria; GFR <60 ml/min/1.73 m2 (CFR categories C3a-C5).

SECONDARY OUTCOMES:
1. Frequency of microalbuminuria, proteinuria, reduced glomerular filtration rate (GFR <60 ml/min/1.73 m²) and other markers of kidney damage in patients with arterial hypertension. | 16 months
  1. Frequency of microalbuminuria, proteinuria, reduced glomerular filtration rate (GFR <60 ml/min/1.73 m²) and other markers of kidney damage in patients with arterial hypertension.
2. Proportion of patients with various risk factors (age, gender, BMI, bad habits, blood pressure, cardiovascular risks) for the development and progression of CKD in patients with arterial hypertension. | 16 months
  2. Proportion of patients with various risk factors (age, gender, BMI, bad habits, blood pressure, cardiovascular risks) for the development and progression of CKD in patients with arterial hypertension.
3.Proportion of patients with various clinical characteristics, such as: • Average and median duration of AH years • Patients with different stages of AH and categories of cardiovascular risk.• Patients with uncontrolled and resistant hypertension. | 16 months
  3. Proportion of patients with various clinical characteristics, such as:
  * Average and median duration of hypertension, years (from the diagnosis date to Visit 1);
  * Patients with different stages of hypertension (I, II, III) and categories of cardiovascular risk (low, moderate, high, very high).
  * Patients with uncontrolled and resistant hypertension.
4. The proportion of patients taking the following groups of drugs for the treatment of AH before inclusion in the study and during participation in the study: • ACE • Alfa or Beta-blockers; • ARBs •CCB • Diuretics • ARNI• Centrally acting drugs; • MRA. | 16 months
  4. The proportion of patients taking the following groups of drugs for the treatment of hypertension before inclusion in the study and during participation in the study:
  * ACE (angiotensin-converting enzyme) inhibitors;
  * Beta-blockers;
  * ARBs (angiotensin receptor blockers);
  * Calcium channel blockers (CCB);
  * Diuretics (thiazide, thiazide-like, loop);
  * Angiotensin receptor-neprilysin inhibitor (ARNI);
  * Alpha-blockers;
  * Centrally acting drugs;
  * Mineralocorticoid receptor antagonists (MRA).
5. Proportion of patients with: • concomitant CVD and complications of AF/AFL, ventricular arrhythmias; CHD; MI; cerebrovascular diseases; stroke, TIA; • other concomitant diseases (in general and for each disease). | 16 months
  5. Proportion of patients with:
  * concomitant cardiovascular diseases (CVD) and complications of hypertension (atrial fibrillation/atrial flutter (AF/AFL), ventricular arrhythmias; coronary heart disease (CHD); myocardial infarction (MI); cerebrovascular diseases; stroke, transient ischemic attack (TIA);
  * other concomitant diseases (in general and for each disease).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Temirlanovka Village, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/